CLINICAL TRIAL: NCT01405820
Title: A Randomized, Blinded, Parallel-Group, Phase 2 Study Exploring the Safety, Tolerability, and Efficacy of Multiple Regimens of Natalizumab in Adult Subjects With Relapsing Multiple Sclerosis
Brief Title: Exploratory Study of the Safety, Tolerability and Efficacy of Multiple Regimens of Natalizumab in Adult Participants With Relapsing Multiple Sclerosis (MS)
Acronym: REFINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101MS206; 2010-024000-10 (EudraCT Number)
Record Dates: First submitted 2011-07-14; First posted 2011-07-29 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Natalizumab 300 mg Intravenous (IV) Every 4 Weeks (Active Comparator): Natalizumab 300 mg IV every 4 weeks for 60 weeks. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
  Interventions: Drug: natalizumab IV
- Natalizumab 300 mg Subcutaneous (SC) Every 4 Weeks (Experimental): Natalizumab 300 mg SC every 4 weeks for 60 weeks. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
  Interventions: Drug: natalizumab IV; Drug: natalizumab SC
- Natalizumab 300 mg IV Every 12 Weeks (Experimental): Natalizumab 300 mg IV every 12 weeks for 60 weeks with matching IV placebo administered during the intervening 4-week periods. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
  Interventions: Drug: natalizumab IV; Drug: IV Placebo
- Natalizumab 300 mg SC Every 12 Weeks (Experimental): Natalizumab 300 mg SC every 12 weeks for 60 weeks with matching SC placebo administered during the intervening 4-week periods. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
  Interventions: Drug: natalizumab IV; Drug: natalizumab SC; Drug: SC Placebo
- Natalizumab 150 mg IV Every 12 Weeks (Experimental): Natalizumab 150 mg IV every 12 weeks for 60 weeks with matching IV placebo administered during the intervening 4-week periods. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
  Interventions: Drug: natalizumab IV; Drug: IV Placebo
- Natalizumab 150 mg SC Every 12 Weeks (Experimental): Natalizumab 150 mg SC every 12 weeks for 60 weeks with matching SC placebo administered during the intervening 4-week periods. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
  Interventions: Drug: natalizumab IV; Drug: natalizumab SC; Drug: SC Placebo

INTERVENTIONS:
Drug: natalizumab IV — natalizumab for IV Infusion
  Other Names: Tysabri; BG00002
Drug: natalizumab SC — natalizumab for Subcutaneous Injection
  Other Names: Tysabri; BG00002
  Arms: Natalizumab 150 mg SC Every 12 Weeks; Natalizumab 300 mg SC Every 12 Weeks; Natalizumab 300 mg Subcutaneous (SC) Every 4 Weeks
Drug: IV Placebo — Intravenous placebo to natalizumab
  Arms: Natalizumab 150 mg IV Every 12 Weeks; Natalizumab 300 mg IV Every 12 Weeks
Drug: SC Placebo — Subcutaneous placebo to natalizumab
  Arms: Natalizumab 150 mg SC Every 12 Weeks; Natalizumab 300 mg SC Every 12 Weeks

SUMMARY:
The primary objective of this study is to explore the effects of multiple regimens of natalizumab on disease activity and safety in participants with relapsing-remitting Multiple Sclerosis (RRMS).

DETAILED DESCRIPTION:
This is a a dose and frequency (but not route of administration) blinded, prospective, randomized, dose-ranging study in patients with RRMS who have received natalizumab for at least 12 months according to the local prescribing guidelines. The study will explore dosing of natalizumab by subcutaneous and intravenous routes. Participants will be randomly assigned to 1 of 6 dosing regimens, blinded to natalizumab dose, but not route, for 60 weeks of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to provide written informed consent
* Subjects of childbearing potential must practice effective contraception during the study
* A documented diagnosis of Relapsing Remitting Multiple Sclerosis (RRMS)
* Free of MS relapse for 12 months prior to randomization
* Treatment with natalizumab for a minimum of 12 months immediately prior to randomization.
* In the 12 months prior to commencing natalizumab, subject must have experienced a minimal level of disease activity as defined by 2 or more documented clinical relapses OR 1 relapse and documented MRI activity, defined by the presence of at least 1 Gd enhancing lesion on MRI, unrelated to the relapse.

Key Exclusion Criteria:

* Known history of Human Immunodeficiency Virus (HIV), hepatitis C and/or hepatitis B virus
* Positive for anti-natalizumab antibodies at screening
* MRI positive for Gd-enhancing lesions at study entry
* Subjects for whom MRI is contraindicated
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic (including diabetes), urologic, pulmonary, neurologic (except for RRMS), dermatologic, psychiatric, renal, or other major disease
* History of malignant disease, including solid tumors and hematologic malignancies (with the exception of cured basal cell and squamous cell carcinomas of the skin)
* History of transplantation or any anti-rejection therapy
* History of severe allergic or anaphylactic reactions or known hypersensitivity to any drug
* A clinically significant infectious illness within 30 days prior to screening or progressive multifocal leukoencephalopathy (PML) or other opportunistic infections at any time
* Signs or symptoms suggestive of any serious infection, based on medical history, physical examination or laboratory testing

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (64):
- Belgium (4):
  - Research Site, Brasschaat
  - Research Site, Liège
  - Research Site, Overpelt
  - Research Site, Wilrijk
- France (11):
  - Research Site, Amiens
  - Research Site, Besançon
  - Research Site, Bron
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (21):
  - Research Site, Andernach
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Dresden
  - Research Site, Emmendingen
  - Research Site, Erbach im Odenwald
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Neuburg am Inn
  - Research Site, Regensburg
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Wermsdorf
- Italy (18):
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Cefalù
  - Research Site, Chieti
  - Research Site, Florence
  - Research Site, Gallarate
  - Research Site, L’Aquila
  - Research Site, Milan
  - Research Site, Montichiari
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Pozzilli
  - Research Site, Roma
  - Research Site, Sassari
  - Research Site, Torino
- Spain (10):
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Girona
  - Research Site, Lleida
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Seville

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four of the 6 arms in the Randomized Treatment Period (the 'every 12 weeks' arms) were closed prematurely. Participants who completed randomized treatment, met rescue criteria, or were impacted by arm closure (and met rescue criteria) were eligible to enroll in the open-label treatment period.
Period: Randomized Treatment Period
Arm/Group | Natalizumab 300 mg Intravenous (IV) Every 4 Weeks | Natalizumab 300 mg Subcutaneous (SC) Every 4 Weeks | Natalizumab 300 mg IV Every 12 Weeks | Natalizumab 300 mg SC Every 12 Weeks | Natalizumab 150 mg IV Every 12 Weeks | Natalizumab 150 mg SC Every 12 Weeks
Started | 54 | 45 | 52 | 54 | 47 | 38
Safety Population | 54 | 45 | 52 | 53 (1 participant did not receive any study medication.) | 47 | 38
Completed | 43 | 35 | 9 | 3 | 2 | 1
Not Completed | 11 | 10 | 43 | 51 | 45 | 37
Not completed — Adverse Event | 3 | 3 | 3 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 6 | 2 | 2 | 2 | 0 | 0
Not completed — Other | 2 | 2 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Rescue | 0 | 1 | 13 | 10 | 8 | 8
Not completed — Incorrect Study Treatment | 0 | 0 | 3 | 0 | 2 | 0
Not completed — Treatment Arm Closed | 0 | 0 | 20 | 36 | 33 | 28
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrew Prior to Dosing | 0 | 0 | 0 | 1 | 0 | 0
Period: Open-Label Treatment Period
Arm/Group | Natalizumab 300 mg Intravenous (IV) Every 4 Weeks | Natalizumab 300 mg Subcutaneous (SC) Every 4 Weeks | Natalizumab 300 mg IV Every 12 Weeks | Natalizumab 300 mg SC Every 12 Weeks | Natalizumab 150 mg IV Every 12 Weeks | Natalizumab 150 mg SC Every 12 Weeks
Started | 44 (1 participant discontinued randomized period due to an adverse event but entered open-label period.) | 35 | 42 | 42 | 42 | 32
Completed | 40 | 33 | 39 | 37 | 40 | 30
Not Completed | 4 | 2 | 3 | 5 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1 | 0 | 1
Not completed — Other | 1 | 1 | 1 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Period: Natalizumab 300 mg IV Every 4 Weeks: Natalizumab 300 mg IV every 4 weeks for 60 weeks.
- Randomized Period: Natalizumab 300 mg SC Every 4 Weeks: Natalizumab 300 mg SC every 4 weeks for 60 weeks.
- Randomized Period: Natalizumab 300 mg IV Every 12 Weeks: Natalizumab 300 mg IV every 12 weeks for 60 weeks with matching IV placebo administered during the intervening 4-week periods.
- Randomized Period: Natalizumab 300 mg SC Every 12 Weeks: Natalizumab 300 mg SC every 12 weeks for 60 weeks with matching SC placebo administered during the intervening 4-week periods.
- Randomized Period: Natalizumab 150 mg IV Every 12 Weeks: Natalizumab 150 mg IV every 12 weeks for 60 weeks with matching IV placebo administered during the intervening 4-week periods.
- Randomized Period: Natalizumab 150 mg SC Every 12 Weeks: Natalizumab 150 mg SC every 12 weeks for 60 weeks with matching SC placebo administered during the intervening 4-week periods.
- Total: Total of all reporting groups
Arm/Group | Randomized Period: Natalizumab 300 mg IV Every 4 Weeks | Randomized Period: Natalizumab 300 mg SC Every 4 Weeks | Randomized Period: Natalizumab 300 mg IV Every 12 Weeks | Randomized Period: Natalizumab 300 mg SC Every 12 Weeks | Randomized Period: Natalizumab 150 mg IV Every 12 Weeks | Randomized Period: Natalizumab 150 mg SC Every 12 Weeks | Total
Number analyzed (Participants) | 54 | 45 | 52 | 54 | 47 | 38 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (7.84) | 36.3 (8.92) | 38.7 (8.43) | 38.7 (7.85) | 38.7 (8.61) | 36.0 (9.03) | 37.9 (8.41)
Age, Customized [Number; unit: participants]
  18 to 19 years | 0 | 1 | 0 | 0 | 0 | 0 | 1
  20 to 29 years | 7 | 11 | 7 | 7 | 5 | 11 | 48
  30 to 39 years | 22 | 15 | 21 | 24 | 21 | 14 | 117
  40 to 49 years | 20 | 16 | 17 | 17 | 16 | 9 | 95
  50 to 56 years | 5 | 2 | 7 | 6 | 5 | 4 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 29 | 37 | 41 | 34 | 24 | 204
  Male | 15 | 16 | 15 | 13 | 13 | 14 | 86

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Combined Unique Active Lesions
Description: Cumulative number of combined unique active lesions (sum of the number of new gadolinium (Gd)-enhancing lesions and new or newly enlarging T2 hyperintense lesions not associated with Gd-enhancement on T1 weighted scans) based on brain magnetic resonance imaging (MRI) scans Up to Week 60.
Time Frame: Up to Week 60
Population: Modified intent-to-treat (mITT) population: all randomized participants who received at least 1 dose of study drug, had at least 1 efficacy assessment, and had no statistical protocol deviations.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Randomized Period: Natalizumab 300 mg IV Every 4 Weeks | Randomized Period: Natalizumab 300 mg SC Every 4 Weeks | Randomized Period: Natalizumab 300 mg IV Every 12 Weeks | Randomized Period: Natalizumab 300 mg SC Every 12 Weeks | Randomized Period: Natalizumab 150 mg IV Every 12 Weeks | Randomized Period: Natalizumab 150 mg SC Every 12 Weeks
Number analyzed (Participants) | 52 | 44 | 45 | 50 | 35 | 32
lesions | 0.23 (1.262) | 0.02 (0.151) | 3.84 (8.054) | 3.08 (8.216) | 6.09 (15.424) | 6.44 (11.285)

ADVERSE EVENTS:
Time Frame: AEs were analyzed during the randomized and open-label (OL) periods separately. Randomized period: AEs, after 1st randomized dose on Day 0 and prior to OL infusion of natalizumab at Week 60 (±5 days); SAEs also between Screening and dosing on Day 0.
Description: OL period: on or after OL infusion of natalizumab at Week 60 through to Week 72 (±2 weeks). If participant did not receive natalizumab infusions during the OL period (Week 60 to Week 72), all events with an onset date after Day 0 were considered as occurring during the randomized treatment period. AE data is presented for the Safety Population.
Groups:
- Open-label Period: Natalizumab 300 mg IV Every 4 Weeks: Natalizumab 300 mg IV every 4 weeks for 60 weeks. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
- Open-label Period: Natalizumab 300 mg SC Every 4 Weeks: Natalizumab 300 mg SC every 4 weeks for 60 weeks. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
- Open-label Period: Natalizumab 300 mg IV Every 12 Weeks: Natalizumab 300 mg IV every 12 weeks for 60 weeks with matching IV placebo administered during the intervening 4-week periods. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
- Open-label Period: Natalizumab 300 mg SC Every 12 Weeks: Natalizumab 300 mg SC every 12 weeks for 60 weeks with matching SC placebo administered during the intervening 4-week periods. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
- Open-label Period: Natalizumab 150 mg IV Every 12 Weeks: Natalizumab 150 mg IV every 12 weeks for 60 weeks with matching IV placebo administered during the intervening 4-week periods. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
- Open-label Period: Natalizumab 150 mg SC Every 12 Weeks: Natalizumab 150 mg SC every 12 weeks for 60 weeks with matching SC placebo administered during the intervening 4-week periods. Open-label natalizumab treatment 300 mg IV at Weeks 60, 64, and 68.
Arm/Group | Randomized Period: Natalizumab 300 mg IV Every 4 Weeks | Randomized Period: Natalizumab 300 mg SC Every 4 Weeks | Randomized Period: Natalizumab 300 mg IV Every 12 Weeks | Randomized Period: Natalizumab 300 mg SC Every 12 Weeks | Randomized Period: Natalizumab 150 mg IV Every 12 Weeks | Randomized Period: Natalizumab 150 mg SC Every 12 Weeks | Open-label Period: Natalizumab 300 mg IV Every 4 Weeks | Open-label Period: Natalizumab 300 mg SC Every 4 Weeks | Open-label Period: Natalizumab 300 mg IV Every 12 Weeks | Open-label Period: Natalizumab 300 mg SC Every 12 Weeks | Open-label Period: Natalizumab 150 mg IV Every 12 Weeks | Open-label Period: Natalizumab 150 mg SC Every 12 Weeks
Serious Adverse Events (participants affected / at risk) | 7/54 | 4/45 | 4/52 | 3/53 | 4/47 | 1/38 | 0/44 | 1/35 | 0/42 | 1/42 | 1/42 | 2/32
Other Adverse Events (participants affected / at risk) | 40/54 | 31/45 | 31/52 | 34/53 | 31/47 | 17/38 | 2/44 | 4/35 | 2/42 | 0/42 | 4/42 | 6/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Period: Natalizumab 300 mg IV Every 4 Weeks (N=54) | Randomized Period: Natalizumab 300 mg SC Every 4 Weeks (N=45) | Randomized Period: Natalizumab 300 mg IV Every 12 Weeks (N=52) | Randomized Period: Natalizumab 300 mg SC Every 12 Weeks (N=53) | Randomized Period: Natalizumab 150 mg IV Every 12 Weeks (N=47) | Randomized Period: Natalizumab 150 mg SC Every 12 Weeks (N=38) | Open-label Period: Natalizumab 300 mg IV Every 4 Weeks (N=44) | Open-label Period: Natalizumab 300 mg SC Every 4 Weeks (N=35) | Open-label Period: Natalizumab 300 mg IV Every 12 Weeks (N=42) | Open-label Period: Natalizumab 300 mg SC Every 12 Weeks (N=42) | Open-label Period: Natalizumab 150 mg IV Every 12 Weeks (N=42) | Open-label Period: Natalizumab 150 mg SC Every 12 Weeks (N=32)
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis Enteroviral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Carcinoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bipolar I Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological Gambling (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Automatic Bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nuclear Magnetic Resonance Imaging Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Period: Natalizumab 300 mg IV Every 4 Weeks (N=54) | Randomized Period: Natalizumab 300 mg SC Every 4 Weeks (N=45) | Randomized Period: Natalizumab 300 mg IV Every 12 Weeks (N=52) | Randomized Period: Natalizumab 300 mg SC Every 12 Weeks (N=53) | Randomized Period: Natalizumab 150 mg IV Every 12 Weeks (N=47) | Randomized Period: Natalizumab 150 mg SC Every 12 Weeks (N=38) | Open-label Period: Natalizumab 300 mg IV Every 4 Weeks (N=44) | Open-label Period: Natalizumab 300 mg SC Every 4 Weeks (N=35) | Open-label Period: Natalizumab 300 mg IV Every 12 Weeks (N=42) | Open-label Period: Natalizumab 300 mg SC Every 12 Weeks (N=42) | Open-label Period: Natalizumab 150 mg IV Every 12 Weeks (N=42) | Open-label Period: Natalizumab 150 mg SC Every 12 Weeks (N=32)
Nasopharyngitis (Infections and infestations) | 13 | 8 | 8 | 9 | 8 | 4 | 2 | 1 | 1 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 8 | 5 | 3 | 4 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 4 | 2 | 1 | 2 | 8 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Pharyngitis (Infections and infestations) | 3 | 1 | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 3 | 0 | 4 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 3 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 4 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 8 | 6 | 13 | 17 | 12 | 5 | 0 | 0 | 1 | 0 | 3 | 2
Headache (Nervous system disorders) | 4 | 9 | 7 | 5 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 6 | 4 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Pain (General disorders) | 0 | 1 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nuclear Magnetic Resonance Imaging Abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.